CLINICAL TRIAL: NCT07193485
Title: Efficacy of Buteyko Breathing in Seniors With Chronic Eustachian Tube Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-36
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): twenty seniors with Eustachian tube dysfunction (chronic obstructive form) will bein group I and this group will take usual care (budesonide spray in nose in 64 microgram concentration one time per day plus the intake of a tablet two times daily containing containing 20-mg contration of pseudoephedrine hydrochloride and 5-mg concentration of loratadine) for 2 weeks. Also, group I will aslo receive 30-min Buteyko breathing two times daily for 14 weeks.
  Interventions: Other: Buteyko breathing
- group number 2 (Active Comparator): Twenty seniors with Eustachian tube dysfunction (chronic obstructive form) will be ranomized to group II oand this group will take usual care (budesonide spray in nose in 64 microgram concentration one time per day plus the intake of a tablet two times daily containing containing 20-mg contration of pseudoephedrine hydrochloride and 5-mg concentration of loratadine) for 2 weeks.
  Interventions: Other: usual care

INTERVENTIONS:
Other: Buteyko breathing — twenty seniors with Eustachian tube dysfunction (chronic obstructive form) will be ranomized to group I and this group will take usual care (budesonide spray in nose in 64 microgram concentration one time per day plus the intake of a tablet two times daily containing containing 20-mg contration of pseudoephedrine hydrochloride and 5-mg concentration of loratadine) for 2 weeks. Also, group I will aslo receive 30-min Buteyko breathing two times daily for 14 weeks.
  Arms: group number 1
Other: usual care — twenty seniors with Eustachian tube dysfunction (chronic obstructive form) will be ranomized to group II and this group will take usual care (budesonide spray in nose in 64 microgram concentration one time per day plus the intake of a tablet two times daily containing containing 20-mg contration of pseudoephedrine hydrochloride and 5-mg concentration of loratadine) for 2 weeks.
  Arms: group number 2

SUMMARY:
Eustachian tube dysfunction is distressing probelm. drugs usually are not effective. compelemtary tehrapies like Buteyko breathing may be effective

DETAILED DESCRIPTION:
forty seniors with Eustachian tube dysfunction (chronic obstructive form) will be ranomized to group I or group II. the group enroled 20 seniors. both groups wil take usual care (budesonide spray in nose in 64 microgram concentration one time per day plus the intake of a tablet two times daily containing containing 20-mg contration of pseudoephedrine hydrochloride and 5-mg concentration of loratadine) for 2 weeks. group I will aslo receive 30-min Buteyko breathing two times daily for 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eustachian Tube Dysfunction (chronic obstructive form)
* unilateral ear affetion
* senior patients
* chronci affection more than 3 months

Exclusion Criteria:

* obesity
* cardiac probelms repsiratory problems

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Eustachian Tube Dysfunction Questionnaire | it will be measured after 2 weeks
  it will be used to asses symptoms of Eustachian Tube Dysfunction

SECONDARY OUTCOMES:
systolic blood pressure | it will be measured after 2 weeks
  it will be measured manually by manual sphygmomanometer
diastolic blood pressure | it will be measured after 2 weeks
  it will be measured manually by manual sphygmomanometer
respiratory rate | it will be measured after 2 weeks
  it will assess breath number per minute
pulse rate | it will be measured after 2 weeks
  it will assess pulse number per minute from radial artery
patient health questionnaire | it will be measured after 2 weeks
  it will assess depression in patients
state trait anxiety inventory | it will be measured after 2 weeks
  it will assess trait anxiety in patients
perceived stress scale | it will be measured after 2 weeks
  it will assess stress in patients
short form 36 questionnaire | it will be measured after 2 weeks
  it will assess quality of life in patients
profile of mood satus | it will be measured after 2 weeks
  it will assess mood in patients
percenatge of tympanometry (type C) | it will be measured after 2 weeks
  it will assess percenatge of type c tympanometry

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Dokki, Giza Governorate, Egypt